CLINICAL TRIAL: NCT04233606
Title: Influence of Osmotic Stimulation of Vasopressin on Autonomic Function
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the university and is no longer in a full time employment role
Sponsor: University of North Carolina, Greensboro (Other)
Responsible Party: Principal Investigator, William Adams, Assistant Professor, University of North Carolina, Greensboro
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20-0206
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Water Stress; Body Water Dehydration
Keywords: Vasopressin; Heart Rate Variability; Cardiovascular Function; Autonomic Function
MeSH Terms: conditions — Dehydration; Diabetes Insipidus | interventions — Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants will complete two trials under two different hydration states: isovolemic increase in plasma osmolality and isovolemic control (maintain normal plasma osmolality)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Participants will be infused with normal (0.9% NaCL) saline for a 120 minute period.
  Interventions: Other: Normal Saline
- Hypertonic Saline (Experimental): Participants will be infused with hypertonic (3% NaCL) saline for a 120 minute period.
  Interventions: Other: Hypertonic Saline

INTERVENTIONS:
Other: Hypertonic Saline — Infusion of hypertonic saline to induce an osmotic secretion of the hormone vasopressin
  Arms: Hypertonic Saline
Other: Normal Saline — Infusion of normal saline to inhibit the secretion of the hormone vasopressin
  Arms: Control

SUMMARY:
The regulation of total body water that defines human hydration status is a complex and dynamic process. Current methods of assessing hydration status (e.g. hematologic and urinary analyses) lack the ability to track changes in hydration status in real-time due to whole-body homeostatic physiologic processes required to maintain central pressure and cardiovascular function. This project will address this problem by assessing the relationship between autonomic function (measured using heart rate variability), a brain-derived process that regulates cardiovascular function, and changes in the hydration-mediated hormone vasopressin.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between the ages of 18 - 35

Exclusion Criteria:

* 1) evidence of clinically relevant diseases that may alter body water regulation (e.g., diabetes, kidney disease, metabolic disorders, cardiovascular disease, and other potential fluid balance covariates such as habitual use of non-steroidal anti-inflammatory drugs or serotonin reuptake inhibitors,

  2) previous surgery on the digestive tract that may impair the body's ability to normally regulate body water,

  3) regular drug treatment within the previous 15 days,

  4) actively attempting to gain or lose body weight,

  5) For female participants, testing will take place during the early follicular phase of their menstrual cycle (days 1-8) to maintain consistency in the hydration status measures as total body water fluctuates over the course of the menstrual cycle. Females who are currently using contraceptives (e.g., IUD) that limit the number of menstrual cycles occurring in a given year will be excluded from this study to ensure accuracy in the testing periods for this study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in autonomic function | 0, 15, 30, 45, 60, 75, 90, 105, 120 minutes of saline infusion period
  Changes in parasympathetic and sympathetic tone as measured by heart rate variability

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina at Greensboro, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No